CLINICAL TRIAL: NCT06882369
Title: Efficacy Of Transversus Abdominis Plane Block , Intrathecal Morphine Or Their Combination For Post Operative Analgesia Following Total Abdominal Hysterectomy.
Brief Title: TAP Block , Intrathecal Morphine Or Their Combination For Post Operative Analgesia Following TAH
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Islam Ahmed Bakr Mohammed, lecturer, Minia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAP vs. morphine vs. both
Record Dates: First submitted 2025-03-07; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Post-operative Pain Management
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TAP block (Active Comparator): Bilateral ultrasound-guided TAP block with 20 mL of 0.25% plain bupivacaine on each side of the abdomen at the end of surgery.
  Interventions: Procedure: TAP Block; Drug: spinal anesthesia
- Intrathecal Morphine (Active Comparator): Intrathecal injection of 100 µg morphine plus 20 mg hyperbaric bupivacaine (in spinal anesthesia).
  Interventions: Drug: Intrathecal morphine injection; Drug: spinal anesthesia
- Combined (Active Comparator): Intrathecal injection of 50 µg morphine plus 20 mg hyperbaric bupivacaine combined with bilateral ultrasound-guided TAP block using 20 mL of 0.25% plain bupivacaine on each side of the abdomen at the end of surgery.
  Interventions: Procedure: TAP Block; Drug: Intrathecal morphine injection; Drug: spinal anesthesia

INTERVENTIONS:
Procedure: TAP Block — The transabdominal plane (TAP) block is a regional anesthesia technique used for postoperative pain management in abdominal wall procedures, providing somatic analgesia to the anterior and lateral abdominal walls
  Arms: Combined; TAP block
Drug: Intrathecal morphine injection — Intrathecal injection of morphine plus 20 mg hyperbaric bupivacaine in spinal anesthesia
  Arms: Combined; Intrathecal Morphine
Drug: spinal anesthesia — intrathecal injection of bupivacaine

SUMMARY:
This randomized controlled clinical trial designed to evaluate the efficacy of transversus abdominis plane (TAP) block, intrathecal morphine, or their combination in postoperative pain relief, as assessed by time to first analgesic request, pain scores, total postoperative analgesic consumption, time of ambulation, complications and hemodynamics following total abdominal hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 30 to 70 years.
* Elective total abdominal hysterectomy.
* ASA physical status I or II.
* Willingness to provide informed consent.

Exclusion Criteria:

* Refusal of the block.
* Allergy to study medications.
* Preexisting coagulation disorders.
* Local infection at the site of needle insertion.
* Uncontrolled respiratory or cardiac disorders.
* Impaired kidney or liver function.

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Time to first analgesic request | 24 hours
  Time (in hours) until the patient demand additional analgesia.

SECONDARY OUTCOMES:
Total analgesic consumption | 24 hours
  Cumulative postoperative analgesic consumption
Time to ambulation | 24 hours
  Time (in hours) from arrival in the PACU until the patient was able to walk.
complications | 24 hours
  Incidence of nausea, vomiting, pruritus, respiratory depression, hematoma, infection or hemodynamic instability

CONTACTS AND LOCATIONS:
Overall Officials: sohair Adeeb, assist.prof., Principal Investigator — Minia University, faculty of medicine
Locations (1):
- Faculty of Medicine, Minia University, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No